CLINICAL TRIAL: NCT05796453
Title: Long-term Evaluation of Safety and Performance of Clareon Presbyopia-Correcting Intraocular Lenses (IOLs)
Brief Title: Post Market Clinical Follow-up (PMCF) Study of Clareon Vivity & Clareon PanOptix
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ILE632-I001
Record Dates: First submitted 2023-03-22; First posted 2023-04-03 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Aphakia; Astigmatism; Presbyopia
Keywords: Cataract surgery
MeSH Terms: conditions — Aphakia; Astigmatism; Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Clareon Vivity IOL - Non Toric (Experimental): Implantation with Clareon Vivity IOLs in both eyes 3-6 months prior to enrollment, with at least one of the eyes implanted with a non-toric Clareon Vivity IOL.
  Interventions: Device: Clareon Vivity IOL - Non Toric
- Clareon Vivity IOL - Toric (Experimental): Implantation with Clareon Vivity IOLs in both eyes 3-6 months prior to enrollment, with at least one of the eyes implanted with a toric Clareon Vivity IOL.
  Interventions: Device: Clareon Vivity IOL - Toric
- Clareon PanOptix IOL - Non Toric (Experimental): Implantation with Clareon PanOptix IOLs in both eyes 3-6 months prior to enrollment, with at least one of the eyes implanted with a non-toric Clareon PanOptix IOL.
  Interventions: Device: Clareon PanOptix Trifocal IOL - Non Toric
- Clareon PanOptix IOL - Toric (Experimental): Implantation with Clareon PanOptix IOLs in both eyes 3-6 months prior to enrollment, with at least one of the eyes implanted with a toric Clareon PanOptix IOL.
  Interventions: Device: Clareon PanOptix Trifocal IOL - Toric

INTERVENTIONS:
Device: Clareon Vivity IOL - Non Toric — Spherical extended vision IOL implanted in the capsular bag of the eye for the visual correction of aphakia in adult patients with less than 1.00 diopter of preoperative corneal astigmatism in whom a cataractous lens has been removed.
  Other Names: Models CNWET0, CCWET0
  Arms: Clareon Vivity IOL - Non Toric
Device: Clareon Vivity IOL - Toric — Toric extended vision IOL implanted in the capsular bag of the eye for the visual correction of aphakia and for reduction of residual refractive astigmatism in adult patients in whom a cataractous lens has been removed.
  Other Names: Models CNWET2, CNWET3, CNWET4, CNWET5, CNWET6, CCWET-2, CCWET3, CCWET4, CCWET3, CCWET3-T6
  Arms: Clareon Vivity IOL - Toric
Device: Clareon PanOptix Trifocal IOL - Non Toric — Spherical trifocal IOL implanted in the capsular bag of the eye for the visual correction of aphakia in adult patients with less than 1.00 diopter of preoperative corneal astigmatism in whom a cataractous lens has been removed.
  Other Names: Model CNWTT0, CCWTT2
  Arms: Clareon PanOptix IOL - Non Toric
Device: Clareon PanOptix Trifocal IOL - Toric — Toric trifocal IOL implanted in the capsular bag of the eye for the visual correction of aphakia and for reduction of residual refractive astigmatism in adult patients in whom a cataractous lens has been removed.
  Other Names: Models CNWTT2, CNWTT3, CNWTT4, CNWTT5, CNWTT6, CCWTT2, CCWTT3, CCWTT4, CCWTT5, and CCWTT6
  Arms: Clareon PanOptix IOL - Toric

SUMMARY:
The purpose of this Post-Market Clinical Follow-up study is to describe the long-term safety and performance of the Clareon Vivity and Vivity Toric and Clareon PanOptix and PanOptix Toric IOLs.

DETAILED DESCRIPTION:
Subjects will be recruited from a population that has already undergone lens implantation. Retrospective data will be collected from the pre-operative and surgical visits and any safety outcomes reported prior to enrollment. Prospective data will be collected from time of study enrollment through the Year 3 follow-up visit.

ELIGIBILITY:
Key Inclusion Criteria:

* Subject or legally authorized representative must be able to understand and sign an approved Informed Consent Form.
* Subject must have had bilateral implantation of Clareon Vivity, Clareon Vivity Toric, Clareon PanOptix, or Clareon PanOptix Toric IOLs between 3-6 months prior to enrollment.
* Subject must have a documented medical history and required pre-operative baseline information available for retrospective data collection.
* Other protocol-defined inclusion criteria may apply.

Key Exclusion Criteria:

* Subject is currently participating in another investigational drug or device study.
* Subject has had corneal refractive surgery after Clareon Vivity, Clareon Vivity Toric, Clareon PanOptix, or Clareon PanOptix Toric IOL implantation.
* Subject is pregnant at the time of enrollment.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Actual)
Dates: Start 2023-09-19 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Mean Binocular Best Corrected Distance Visual Acuity (BCDVA) at each prospective visit | Up to Year 3
  BCDVA will be assessed at a distance of 4 meters using letter charts and recorded in logarithm Minimum Angle of Resolution (logMAR).
Rate of Adverse Events | Up to Year 3
  Protocol-specified ocular adverse events will be assessed at each prospective visit and include the following:
  * Cystoid Macular Edema (CME)
  * Hypopyon
  * Endophthalmitis
  * Lens dislocation
  * Pupillary Block
  * Retinal Detachment
  * Secondary Surgical Interventions (Explantation/exchange/repositioning)
Rate of Device Deficiencies | Up to Year 3
  Device deficiencies will be assessed at each prospective visit. Examples include the following:
  * Failure to meet product specifications (e.g., incorrect IOL power)
  * IOL defect
  * Broken IOL optic
  * Broken IOL haptic
  * Scratched IOL optic
  * Unsealed device packaging
  * Suspected product contamination
  * Lack of performance

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Surgical, Study Director — Alcon Research, LLC
Locations (7):
- United States (6):
  - Wolstan & Goldberg Eye Associates, Torrance, California
  - Levenson Eye Associates, Jacksonville, Florida
  - Eye Surgeons of CNY, Liverpool, New York
  - Tulsa Ophthalmology, Tulsa, Oklahoma
  - Chu Eye Institute, Fort Worth, Texas
  - The Eye Institute of Utah, Salt Lake City, Utah
- Centro Oftalmologico Metropolitano, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No